CLINICAL TRIAL: NCT01887418
Title: 3 Arm Open-label Randomized Multidose Study of Pharmacokinetics, Safety & Tolerability of Testosterone Enanthate Administered Subcutaneously Via an Auto-injector Device or Intramuscular Testosterone Enanthate in Hypogonadal Adult Males
Brief Title: Pharmacokinetic Study of Testosterone Enanthate
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Antares Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QST-13-002
Record Dates: First submitted 2013-06-17; First posted 2013-06-26 (Estimated); Results first posted 2015-10-21 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2017-12

CONDITIONS: Hypogonadism
Keywords: Hypogonadism; Testosterone enanthate
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone; testosterone enanthate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- QuickShot™ - 100 mg Treatment A (Experimental): QuickShot™Testosterone - Auto-injector device for SC use
  Interventions: Drug: QuickShot™ - 100 mg Treatment A
- QuickShot™ - 50 mg Treatment B (Experimental): QuickShot™Testosterone- Auto-injector device for SC use
  Interventions: Drug: QuickShot™ - 50 mg Treatment B
- Delatestryl 200 mg IM Treatment C (Active Comparator): Commercially available Testosterone enanthate 200 mg IM dosage - 'standard of care' arm for reference
  Interventions: Drug: Delatestryl 200 mg IM Treatment C

INTERVENTIONS:
Drug: QuickShot™ - 50 mg Treatment B — QuickShot™ for the delivery of testosterone
  Other Names: Testosterone; Testosterone enanthate
  Arms: QuickShot™ - 50 mg Treatment B
Drug: QuickShot™ - 100 mg Treatment A — QuickShot™ for the delivery of testosterone
  Other Names: Testosterone; Testosterone enanthate
  Arms: QuickShot™ - 100 mg Treatment A
Drug: Delatestryl 200 mg IM Treatment C — Standard of care
  Other Names: Testosterone; Testosterone enanthate
  Arms: Delatestryl 200 mg IM Treatment C

SUMMARY:
Relative Bioavailability and Safety comparison of 3 formulations of Testosterone Enanthate.

DETAILED DESCRIPTION:
Standard Pharmacokinetic (PK) analyses of data for serum testosterone were done. Cmax, Area Under Curve (AUC), and Cavg were used for the comparison of relative bioavailability of the treatments and reference arm.

Safety comparisons were based upon the occurrence, severity and rate of treatment emergent adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Adult males aged 18 to 75 with a documented diagnosis of hypogonadism

Exclusion Criteria:

* Normal testosterone levels
* Subjects with any clinically significant medical condition which, in the opinion of the Investigator, would make the subject an unsuitable candidate for enrollment in the study

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Bedel, MD, Principal Investigator — Prestige Clinical Research
Locations (1):
- Mens Health Boston, Brookline, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened at 10 sites in USA. In total, 39 eligible subjects were enrolled and received study medication (investigational SC QST or IM RLD): 14 subjects in 50 mg SC QST arm, 15 subjects in 100 mg SC QST arm and 10 subjects in 200 mg IM RLD arm.
Pre-assignment Details: Eligible patients were randomized to receive SC 50mg (Treatment B) or SC 100mg (Treatment A) QST and the subject who were on IM testosterone replacement therapy, received IM TE RLD (Treatment C).
Groups:
- QuickShot™ - 100 mg Treatment A: QuickShot™ - Auto-injector device for SC use
  QuickShot™ - 100 mg Treatment A: QuickShot™ for the delivery of testosterone once a week
- QuickShot™ - 50 mg Treatment B: QuickShot™ - Auto-injector device for SC use
  QuickShot™ - 50 mg Treatment B: QuickShot™ for the delivery of testosterone once a week.
- Delatestryl 200 mg IM Treatment C: Commercially available Testosterone enanthate 200 mg IM dosage - 'standard of care' arm for reference
  Delatestryl 200 mg IM Treatment C: injected once only
Period: Overall Study
Arm/Group | QuickShot™ - 100 mg Treatment A | QuickShot™ - 50 mg Treatment B | Delatestryl 200 mg IM Treatment C
Started | 15 | 14 | 10
Completed | 15 | 14 | 9
Not Completed | 0 | 0 | 1
Not completed — Travelling difficulties | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Population (39 subjects) was all randomized subjects who received at least 1 dose of investigational product.
  The PK Population (39 subjects) was all subjects from Safety Population who did not have a major protocol deviation that impacted the integrity of PK data and had at least 1 valid post-dose plasma concentration value.
Groups:
- QuickShot™ - 100 mg Treatment A: QuickShot™ - Auto-injector device for SC use
  QuickShot™ - 100 mg Treatment A: QuickShot™ for the delivery of testosterone once a week for 6 weeks
- QuickShot™ - 50 mg Treatment B: QuickShot™ - Auto-injector device for SC use
  QuickShot™ - 50 mg Treatment B: QuickShot™ for the delivery of testosterone once a week for 6 weeks
- Total: Total of all reporting groups
Arm/Group | QuickShot™ - 100 mg Treatment A | QuickShot™ - 50 mg Treatment B | Delatestryl 200 mg IM Treatment C | Total
Number analyzed (Participants) | 15 | 14 | 10 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (12.80) | 54.0 (12.42) | 48.9 (10.94) | 52.9 (12.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 15 | 14 | 10 | 39
Race/Ethnicity, Customized [Number; unit: participants]
  White | 13 | 14 | 8 | 35
  African American | 2 | 0 | 1 | 3
  Multiple | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 15 | 14 | 10 | 39
Body Mass Index (BMI) at screening (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 29.19 (2.87) | 28.51 (2.17) | 29.05 (2.21) | 28.91 (2.43)
Baseline Total Testosterone (TT) (ng/dL) [Mean (Standard Deviation); unit: ng/dL] | 201.50 (71.53) | 214.64 (59.05) | 735.10 (187.96) | 343.04 (256.67)

OUTCOME MEASURES:

1. Secondary Outcome: Number of Patients in the PK Parameter Category
Description: The number of TT Cavg (0-168h) values within the normal range (300-1100 ng/dL) following treatment with SC TE administered via QST or IM TE
Time Frame: 6 weeks
Measure: Number; unit: participants
Groups:
- QuickShot™ - 100 mg Treatment A: QuickShot™ - Auto-injector device for SC use
  QuickShot™ - 100 mg Treatment A: QuickShot™ for the delivery of testosterone
- QuickShot™ - 50 mg Treatment B: QuickShot™ - Auto-injector device for SC use
  QuickShot™ - 50 mg Treatment B: QuickShot™ for the delivery of testosterone
Arm/Group | QuickShot™ - 100 mg Treatment A | QuickShot™ - 50 mg Treatment B | Delatestryl 200 mg IM Treatment C
Number analyzed (Participants) | 15 | 14 | 10
participants | 10 | 12 | 3

2. Primary Outcome: The Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)] of Testosterone Enanthate Formulations at 6 Weeks
Description: The area under the curve from time zero to last quantifiable concentration [AUC (0-t)] of TE administered by SC injection once weekly at doses of 50 mg and 100 mg via the QST
Time Frame: 0, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 and 168 hours post-dose, at 6 Weeks
Population: PK profile of TT obtained at Week 6 of treatment by QST
Measure: Mean (Standard Deviation); unit: ng*hr/dL
Arm/Group | QuickShot™ - 100 mg Treatment A | QuickShot™ - 50 mg Treatment B | Delatestryl 200 mg IM Treatment C
Number analyzed (Participants) | 15 | 14 | 10
ng*hr/dL | 150445.2 (46998.76) | 70955.7 (20815.18) | 278657.9 (168295.52)

3. Primary Outcome: The Maximum Plasma Concentration [Cmax] of Testosterone Enanthate Formulations at 6 Weeks
Description: The maximum observed plasma concentration [Cmax] of TE administered by SC injection once weekly at doses of 50 mg and 100 mg via the QST
Time Frame: 0, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 and 168 hours post-dose, at 6 Weeks
Population: PK profile of TT obtained at Week 6 of treatment by QST
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | QuickShot™ - 100 mg Treatment A | QuickShot™ - 50 mg Treatment B | Delatestryl 200 mg IM Treatment C
Number analyzed (Participants) | 15 | 14 | 10
ng/dL | 1345.6 (435.63) | 622.4 (129.51) | 261.9 (1310.34)

4. Primary Outcome: The Average Concentration [Cavg] of Testosterone Enanthate Formulations at 6 Weeks
Description: The average concentration [Cavg] of TE administered by SC injection once weekly at doses of 50 mg and 100 mg via the QST
Time Frame: 0, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 and 168 hours post-dose, at 6 Weeks
Population: PK profile of TT obtained at Week 6 of treatment by QST
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | QuickShot™ - 100 mg Treatment A | QuickShot™ - 50 mg Treatment B | Delatestryl 200 mg IM Treatment C
Number analyzed (Participants) | 15 | 14 | 10
ng/dL | 895.5 (279.75) | 422.4 (123.90) | 1658.7 (1001.76)

ADVERSE EVENTS:
Time Frame: Adverse events were classified as any adverse events that occurred from Day1 (after screening) to a given treatment period until the subject completed the study. The duration of the study participation for subjects was approximately 19 weeks.
Description: The Safety Population was defined as all randomized subjects who received at least 1 dose of investigational product. The safety population was 39 subjects.
Arm/Group | QuickShot™ - 100 mg Treatment A | QuickShot™ - 50 mg Treatment B | Delatestryl 200 mg IM Treatment C
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14 | 0/10
Other Adverse Events (participants affected / at risk) | 7/15 | 6/14 | 0/10
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | QuickShot™ - 100 mg Treatment A (N=15) | QuickShot™ - 50 mg Treatment B (N=14) | Delatestryl 200 mg IM Treatment C (N=10)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site hematoma (General disorders) | 2 (2) | 1 (1) | 0 (0)
Injection site hemorrhage* (General disorders) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Prostatic specific antigen increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less